CLINICAL TRIAL: NCT00707473
Title: Phase II Trial of Induction Therapy With Docetaxel, Cisplatin and Fluorouracil in Previously Untreated Patients With Locally Advanced Squamous Cell Carcinoma and/or Poorly Differentiated Carcinoma of the Nasal Cavity and/or Paranasal Sinuses
Brief Title: Docetaxel, Cisplatin and Fluorouracil in Treating Patients With Previously Untreated Stage II-IV Nasal Cavity and Paranasal Sinus Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0433; NCI-2018-01810 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2007-0433 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma; Nasal Cavity and Paranasal Sinus Poorly Differentiated Carcinoma; Sinonasal Undifferentiated Carcinoma; Stage II Nasal Cavity and Paranasal Sinus Cancer AJCC v8; Stage III Nasal Cavity and Paranasal Sinus Cancer AJCC v8; Stage IVA Nasal Cavity and Paranasal Sinus Cancer AJCC v8; Stage IVB Nasal Cavity and Paranasal Sinus Cancer AJCC v8
MeSH Terms: conditions — Sinonasal undifferentiated carcinoma; Paranasal Sinus Neoplasms | interventions — Carboplatin; Chemoradiotherapy; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Docetaxel; Fluorouracil; dehydroftorafur; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (docetaxel, cisplatin, and fluorouracil) (Experimental): INDUCTION CHEMOTHERAPY: Patients receive docetaxel IV over 1 hour on day 1, cisplatin IV over 30-180 minutes or carboplatin IV on day 1, and fluorouracil IV continuously on days 1-4. Cycles repeat every 3 weeks for up to 2 cycles in the absence of disease progression or unacceptable toxicity.
  Patients who achieve CR or PR receive 1 additional course of treatment and undergo chemoradiotherapy over 6-7 weeks. Patients who have SD or PD to induction therapy, or less than a complete response to chemoradiotherapy undergo surgery and radiation therapy.
  Interventions: Drug: Carboplatin; Other: Chemoradiotherapy; Drug: Cisplatin; Procedure: Definitive Surgical Resection; Drug: Docetaxel; Drug: Fluorouracil; Procedure: Quality-of-Life Assessment; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Other: Chemoradiotherapy — Undergo chemoradiotherapy
  Other Names: chemoradiation
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Definitive Surgical Resection — Undergo surgery
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Procedure: Quality-of-Life Assessment — Correlative studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation

SUMMARY:
This phase II trial studies how well docetaxel, cisplatin and fluorouracil work in treating patients with previously untreated stage II-IV nasal cavity and/or paranasal sinus cancer. Drugs used in chemotherapy, such as docetaxel, cisplatin and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the clinical/radiographic complete and partial response rate after induction chemotherapy with docetaxel, cisplatin and fluorouracil (TPF).

II. To improve local tumor control to 80% at 2 years.

SECONDARY OBJECTIVES I. Disease specific-survival and overall survival rates. II. Organ preservation (orbital, maxillary, cranial) rate. III. Patterns of treatment failure (local, regional, and distant). IV. Acute and late treatment-related toxicity. V. The effect of treatment on Quality of Life with and without surgery (i.e., M. D. Anderson Symptom Inventory [MDASI], M. D. Anderson Dysphagia Inventory [MDADI], Xerostomia Questionnaire, Performance Status Scale for Head & Neck Cancer Patients [PSS-HN], etc.).

VI. To evaluate the effects of induction chemotherapy on biological markers that could serve as surrogates for response and predictors of long-term outcome.

OUTLINE:

INDUCTION CHEMOTHERAPY: Patients receive docetaxel intravenously (IV) over 1 hour on day 1, cisplatin IV over 30-180 minutes or carboplatin IV on day 1, and fluorouracil IV continuously on days 1-4. Cycles repeat every 3 weeks for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

Patients who achieve complete response (CR) or partial response (PR) receive 1 additional course of treatment and undergo chemoradiotherapy over 6-7 weeks. Patients who have stable disease (SD) or progressive disease (PD) to induction therapy, or less than a complete response to chemoradiotherapy undergo surgery and radiation therapy.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 4 months for 1 year and every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed (by a MD Anderson Cancer Center [MDACC] pathologist) cytologic or histological diagnosis of locally advanced squamous cell carcinoma, poorly differentiated carcinoma, or sinonasal undifferentiated carcinoma of the nasal cavity and/or paranasal sinuses.
* Stage II-IV disease; tumor (T) 2-4, node (N) any, metastasis (M) 0. Measurable disease is required with the following criteria: Measurable lesions can be accurately measured, with at least one diameter >= 1.0 cm by spiral computed tomography (CT) scan or magnetic resonance imaging (MRI). Lesions can be bidimensionally measurable or unidimensionally measurable. Every effort should be made to measure lesions in two dimensions. Measurable disease is present if the patient has one or more measurable lesions. Non-measurable lesions/disease are all other lesions, including small lesions (those with measurements < 2.0 cm; or < 1.0 cm with spiral CT).
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1.
* Absolute peripheral granulocyte count (AGC) of >= 1500 cells/mm^3.
* Platelet count of >= 100,000 cells/mm^3.
* Total bilirubin =< upper limit of normal (ULN). If the patient has a history of Gilbert's Syndrome, check direct and indirect bilirubin. If in the judgment of the attending medical oncologist it is safe to treat the patient, the patient will be considered eligible for this criteria.
* Alkaline phosphatase =< 2 x ULN. If in the judgment of the attending medical oncologist it is safe to treat the patient, the patient will be considered eligible for this criteria.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2 x ULN. If in the judgment of the attending medical oncologist it is safe to treat the patient, the patient will be considered eligible for this criteria.
* Hemoglobin >= 10.0g/dL.
* Per MDACC creatinine clearance (CrCl) guidelines, patients must have a creatinine clearance > 50 ml/min determined by 24 hour collection or nomogram
* Patients should have uncontrolled intercurrent illness, which in the opinion of the attending medical oncologist, would render the patient unsuitable for the study (i.e., preclude safe administration of the prescribed chemotherapy treatment).
* Women of child bearing potential (WOCBP) must have a negative serum or urine pregnancy test (i.e., minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]), within 72 hours prior to the start of study treatment. Should a woman become pregnant or suspect she is pregnant while participating in the study, she should inform her treating physician(s) immediately.
* Ability to understand and the willingness to sign a written Informed Consent Document (ICD). In the event that non-English speaking participants are eligible for this study, a short form (if applicable) or an ICD in their language, will be utilized and completed in accordance with the MDACC Policy For Consenting Non-English Speaking Participants.
* Willingness to undergo MDACC Audiology and Ophthalmology Assessment.

Exclusion Criteria:

* Evidence of distant metastases (below the clavicle) by clinical or radiographic measures.
* Pre-existing peripheral neuropathy Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or worse.
* Pre-existing bilateral sensorineural hearing loss at > 90dB at any frequency from 250-8000Hz as assessed by a comprehensive audiometric evaluation for patients receiving cisplatin. This criteria will not apply to patients receiving carboplatin.
* Prior chemotherapy (i.e., as administered strictly for cancer treatment) within the previous 3 years. Use of chemotherapy agents for non-cancer treatment purposes (i.e., arthritis treatment, etc.) are excluded from this criterion.
* Prior radiotherapy to the paranasal sinus region or the upper neck (i.e., prior radiotherapy to another disease site is acceptable).
* Initial surgical resection of the paranasal sinuses or nasal cavity region rendering the patient clinically and radiologically disease free.
* Simultaneous primary invasive cancers or patients currently receiving any other investigational agents at time of study enrollment. Patients may have received investigational agents in the past. No washout time period is required.
* Patients with a past history of malignancy that were treated less than 3 years and have not remained disease free for the past 3 years. (Patients with non metastatic skin cancers will be eligible).
* Men and women of childbearing potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 3 months after the study. Subjects who are men must also agree to use effective contraception. Note: WOCBP must be using an adequate method of contraception throughout the study and for up to 3 months after the study. Adequate methods of contraception will include (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner).
* Women who are pregnant or breastfeeding.
* Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80.
* Patients with a known history of human immunodeficiency virus (HIV).

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-06-16 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical/radiographic complete rate after induction chemotherapy with docetaxel, cisplatin, and fluorouracil | Up to 5 years
Local tumor control to 80% | At 2 years

SECONDARY OUTCOMES:
Disease specific-survival rate | Up to 5 years
Overall survival rate | Up to 5 years
Organ preservation (orbital, maxillary, cranial) rate | Up to 5 years
Patterns of treatment failure (local, regional, and distant) | Up to 5 years
Acute treatment-related toxicity | U to 5 years
Late treatment-related toxicity | Up to 5 years
Quality of Life with and without surgery | Up to 5 years
Biological markers | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Y Hanna, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org